CLINICAL TRIAL: NCT03712215
Title: ELECTRICAL DIAPHRAGMATIC STIMULATION IN PULMONARY FUNCTION OF CRITICAL PATIENTS
Brief Title: STUDY OF ELECTRICAL STIMULATION IN PULMONARY FUNCTION IN INTENSIVE CARE UNIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Metodista de Piracicaba (Other)
Collaborators: Universidade do Estado do Pará (Other)
Responsible Party: Principal Investigator, Rodrigo Santiago Barbosa Rocha, Phd, Principal invastigator, Universidade Metodista de Piracicaba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1.762.021
Record Dates: First submitted 2018-09-03; First posted 2018-10-19 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: Mechanical Ventilation; Electrical Stimulation; Diaphragm; Ventilometry; Physiotherapy
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group 1 (Experimental): synchronized FES mode, according to the parameters based on the Gueddes et al., (1991): current frequency (F) 30 Hz; pulse width (T) 0,4 ms; upload time (Rise) 1s; time of muscle contraction (On time) 1 s; down time (Decay) 2s e muscle relaxation time (Off time) 1 s.
  Interventions: Other: Rehabilitation
- Experimental Group 2 (Experimental): the same apparatus will be used, differing in the parameters that will be based on the studies of Cancelliero et al., (2012) for the EDET procedure, being used in synchronized FES mode, with frequency of 30 Hz; pulse width (T) 0,4 ms, climb (ramp) of 0,7 s (maximum value). The support was of 0.4 s, already standardized and fixed in the apparatus
  Interventions: Other: Rehabilitation
- Control Group (No Intervention): The control group (CG) with the same characteristics of the experimental groups will perform conventional physiotherapy

INTERVENTIONS:
Other: Rehabilitation — diaphragmatic electrical stimulation
  Arms: Experimental Group 1; Experimental Group 2

SUMMARY:
Introduction: The Mechanical Ventilation (MV), a support method used in Intensive Care Units (ICU), reaches approximately 90% of critical patients whose withdrawal process represents 40% of the total time of their use. For this purpose Transcutaneous electrical diaphragmatic stimulation (TEDS), which by means of electrodes placed in motor action points on the phrenic nerve tend to provide improvement of the diaphragm muscle function. Objective: To analyze the effect of two protocols of transcutaneous electrical diaphragmatic stimulation on the ventilatory and cardiorespiratory parameters of critically ill patients. Method: Clinical, longitudinal, prospective, quantitative, single center trial will be performed with 30 (thirty) participants in invasive mechanical ventilatory support, randomly divided into three groups: Experimental Group 1 (GE-1; n = 10) where they will be submitted to the TEDS protocol; Experimental Group 2 (GE-2; n = 10), where they will be submitted to the TEDS protocol based on the studies of Cancelliero et al. (2012); Control Group (GC; n = 10) where they will not be submitted to TEDS. All groups will receive physiotherapeutic care from the staff of the adult ICU of the FHCGV. The interventions will consist of ten sessions of Physical Therapy in each participant in the afternoon shift, for ten consecutive days, 1 time a day. For the TEDS procedure, the Orion TENS II (Orion-SP-Brazil) model will be used, the Wright analogue respirometer (Spire-SP-Brazil) will be used for the minute volume evaluation (V'). The variables of systolic blood pressure (SBP), diastolic blood pressure (DBP), heart rate (HR) and peripheral oxygen saturation (SpO2) will also be monitored in order to verify if the TEDS application interferes with the hemodynamic variables of these patients. The data collected will be linked to Microsoft Office Excel® 2010 software and later transformed into tables and graphs. The information collected will be submitted to statistical analysis through the statistical package SPSS 22.0, applying the descriptive statistics for the characterization of the sample and then selecting the specific tests for the respective variances, adopting a level of significance of p≤0.05 for statistical inferences.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of both sexes aged 60 years and older up to 80 years,
* in invasive MV for more than 48 hours,
* with respiratory drive,
* using MV in the mode of intermittent mandatory synchronized ventilation (VMIS) or (VPS),
* connected to the orotracheal tube or via tracheostomy,
* hemodynamically stable,
* neuromuscular junction of the entire diaphragm,
* absence of sedatives.

Exclusion Criteria:

* presence of pacemaker, hyperthermia (temperature> 38 ° C),
* use of neuromuscular blockers,
* use of thoracic drains, generalized edema,
* cutaneous lesion in the area of intervention with TEDS.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Individuals aged 60 years and older up to 80 years
Enrollment: 30 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Minute volume | From date of randomization until the date of first documented progression, assessed up to 24 months
  For the evaluation of the minute volume will be used Wright analog breathing apparatus. This analysis will occur during the initial evaluation and at the end of each service. For measurement, the ventilometer will be connected to a filter of the brand HMEF UNDIS MEDICAL for adults with extensible trachea of 15 cm, and it is attached directly to the tracheostomy cannula. The patient will remain for a maximum of one minute outside the MV, obstructing the nose with nose clip to thus measure the minute volume spontaneously.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Clínicas Gaspar Viana, Belém, Pará, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Yabek SM, Jarmakani JM. Sinus node dysfunction in children, adolescents, and young adults. Pediatrics. 1978 Apr;61(4):593-8. PMID 662485
- [Result] Wachtel SS, Basrur P, Koo GC. Recessive male-determining genes. Cell. 1978 Sep;15(1):279-81. doi: 10.1016/0092-8674(78)90103-4. PMID 699047
- [Result] Geddes LA, Voorhees WD, Bourland JD, Riscili CE. Optimum stimulus frequency for contracting the inspiratory muscles with chest-surface electrodes to produce artificial respiration. Ann Biomed Eng. 1990;18(1):103-8. doi: 10.1007/BF02368420. PMID 2306029
- [Result] Krymskii LD, Nestaiko GV. [Scanning electron microscopy of vessels in normal and pathologic states]. Vestn Akad Med Nauk SSSR. 1975;(11):71-6. No abstract available. Russian. PMID 775835
- [Result] Arguelles JE, Franatovic Y, Romo-Salas F, Aldrete JA. Intrabiliary pressure changes produced by narcotic drugs and inhalation anesthetics in guinea pigs. Anesth Analg. 1979 Mar-Apr;58(2):120-3. PMID 35040